CLINICAL TRIAL: NCT03899194
Title: Study on the Effect of PRKCB1 Modulating Inflammatory Factors and the Role for Developing Major Depressive Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, Yiru FANG M.D., Ph.D., Director, Shanghai Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 81771465
Record Dates: First submitted 2019-02-21; First posted 2019-04-02 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-04

CONDITIONS: Major Depressive Disorder
Keywords: major depressive disorder; neuroimmunology; PRKCB1 gene; modulation; biomarker
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Fish Oils; Escitalopram

STUDY DESIGN:
Intervention Model Description: group 1: escitalopram group 2: escitalopram + Omega-3 PUFAs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- escitalopram (Active Comparator): Patients will only be treated with escitalopram from the minimum dosage.
  Interventions: Drug: escitalopram
- escitalopram+ fish oil capsules (Experimental): Patients will be treated with escitalopram from the minimum dosage and fish oil capsules according to direction for use.
  Interventions: Dietary Supplement: fish oil capsules

INTERVENTIONS:
Dietary Supplement: fish oil capsules — fish oil capsules(1000mg，EPA 180mg；DHA 120mg)
  Arms: escitalopram+ fish oil capsules
Drug: escitalopram — escitalopram 10-20 mg/d
  Arms: escitalopram

SUMMARY:
Depressive disorder is known as being accompanied with the activation of immune system which could lead to a series of changes including the neuron apoptosis, synapses transmission inhibition and emotional symptoms. The activation of protein kinase C (PKC) can reverse the immune/inflammatory process and restore the neuroplasticity and neurotransmitters transmission. Based on our finding that patients with major depressive disorder (MDD) showed a significantly lower gene expression of PRKCB1, while the PKC activation mediated by PRKCB1, we hypothesize that PRKCB1 contribute to the development of MDD and treatment response by its specific expression in brain, regulating ERBB, Chemokine signaling pathways and PKC activation during the neuroinflammatory process. In the present study, we aim to evaluate and verify the regulation effect of PRKCB1 on the neuroimmune and inflammatory mechanism in depressive disorder by a serious of studies focus on PRKCB1 gene expression modulating process and different downstream biomarkers which associated with PRKCB1 effect, combined with the specified treatment (plus omega-3 poly unsaturated fat acids). This study may provide scientific evidences for using neuroinflammatory biomarkers to diagnose MDD, as well as personalized treatment.

DETAILED DESCRIPTION:
(1）To find out the differences of expression of mRNA, lncRNA, miRNA and proteins of PRKCB1 between patients with depressive disorder and healthy subjects.

(2) Patients with depressive disorders will be randomized into two groups that they will be treated with escitalopram or escitalopram plus Omega-3 PUFAs. To observe the effects of Omega-3 PUFAs on PRKCB1 and related neuroimmune/neuroinflammatory pathway which may improve understanding the relationship between neuroinflammatory regulation and depressive disorder treatment.

ELIGIBILITY:
Inclusion Criteria for patients:

1. Drug-naive or medication free for no less than 4 weeks;
2. 18-60 years old, Han nationality;
3. Junior high school diploma or above;
4. Meeting with the criteria of major depressive disorder in the Diagnostic and Statistical Manual of Mental Disorders (DSM)-IV-TR;
5. Scored 17 or higher on the Hamilton's Depression Scale with 17 items (HAMD-17) and scored 2 or higher for the 2nd item (depressive mood);
6. Written informed consent has been obtained.

Exclusion Criteria for patients:

1. Concurring psychotic disorders;
2. Woman who is pregnant or breast feeding or is planning to get pregnant;
3. Scores 3 or higher on item 3 (suicidal) of HAMD-17;
4. serious allergy or disease of immune system;
5. had anti-inflammatory drug or immunosuppressant in the past 1 month;
6. serious medical or surgical illness or history;
7. had MECT in the past 1 month.

Eligibility Criteria for healthy volunteers:

1. match the patient group in age, gender, education and handedness;
2. no history of psychiatric disorders or debilitating general medical disorders.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 350 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
remission of acute phase | 12th week
  scored 7 or lower on the Hamilton's Depression Scale with 17 items
remission of consolidate and maintenance phase | 12th month
  scored 7 or lower on the Hamilton's Depression Scale with 17 items

CONTACTS AND LOCATIONS:
Overall Officials: Yiru Fang Fang, MD. PhD., Study Chair — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Appleton KM, Voyias PD, Sallis HM, Dawson S, Ness AR, Churchill R, Perry R. Omega-3 fatty acids for depression in adults. Cochrane Database Syst Rev. 2021 Nov 24;11(11):CD004692. doi: 10.1002/14651858.CD004692.pub5. PMID 34817851